CLINICAL TRIAL: NCT03410381
Title: Development of an Algorithm and a Smartphone Application for the Evaluation and Prediction of Suicidal Risk
Brief Title: Ecological Momentary Mental Assessment
Acronym: EMMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Collaborators: University Hospital, Lille (Other); University Hospital, Brest (Other); University Hospital Saint jacques, Besançon (Unknown); University Hospital, Henri Mondor/Albert Chenevier, Créteil (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 9867; 2017-A22108-45 (Other: Agence Nationale de Securité des Médicaments et produist de santé)
Record Dates: First submitted 2017-12-14; First posted 2018-01-25 (Actual); Last update posted 2021-02-05 (Actual); Status verified 2021-01

CONDITIONS: Person at Risk of Suicide
Keywords: Psychiatry; Suicide; Prediction; Smartphone application; Ecological Momentary Assessment
MeSH Terms: conditions — Suicide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Group using the application EMMA (Experimental): Patients with personal history of suicide attempt or with suicidal ideation, will use the application during 6 months. Assessment of the predictive value of the algorithm for suicidal risk, acceptbability and satisfaction
  Interventions: Other: Application EMMA

INTERVENTIONS:
Other: Application EMMA — Emma proposes four types of assessments during 6 months:1) 5 times a day during 3 days, every month (5 minutes): patients can assess their emotions, their thoughts, their behavior and their occurrence context. 2) Weekly (7 minutes): consists of a summary of the week, about their emotions, thoughts, behavior, their relationships (family, work, friends, and their quality of life.3) Monthly (5 minutes): assessment of the usefulness and satisfaction about the application.4) Assessment available at any time An action plan is designed to support the participants, to help them facing difficult emotions and feelings, and to encourage them to ask for help. They can contact a relative or call the psychiatric emergency service directly by clicking on a button.

SUMMARY:
Suicide is a major health problem that causes annually a million death worldwide. Suicide and suicide attempts are preventable.

A history of self-injuries or suicidal attempts are known to be the most important risk factor for death by suicide. Suicidal ideation is also strongly correlated with suicide attempts.

The development of Smartphones applications offers new possibilities for data collection and transmission.

Moreover, the online help function, when a suicidal crisis occurs, is the most effective strategy for prevention of suicidal behavior.

Specific technologies have been developed to analyse behaviors and experiences of patients in a natural environment, in real life.

That is the goal of Ecological Momentary Assessment.

The aim of the study is to develop an algorithm to assess and predict the risk of suicidal event occurrence, in order to detect as soon as possible the signs of suicidal crisis.

EMMA will be the first application in French, meeting the recommendations for health applications, developed by experts on suicidal behavior and in collaboration with patients which aims to predict suicidal risk.

A subsequent study, conducted on a larger population, should allow to validate the predictive algorithm of EMMA.

Long-term goal is to improve the care of patients at risk for suicidal behavior.

DETAILED DESCRIPTION:
100 patients having recently attempted suicide or having suicidal ideation will be recruited. They will be asked to use the application EMMA during 6 months and will be followed up during this period.

An optional qualitative study conducted on 25 patients will allow to evaluate more finely their subjective experience of the use of the application.

Initial visit (inclusion) : clinical, biological and neuropsychological assessment and installation of the application EMMA.

First visit (1st month) and second visit (3rd month) : clinical assessment

Last visit (6th month) : clinical, biological and neuropsychological assessment and optional qualitative interview.

ELIGIBILITY:
Inclusion Criteria:

* Recent suicidal attempt (< 8 days) or suicidal ideation score ≥ 2 (IDSC-30 scale)
* More than 18 years old
* Able to understand nature, aims, and methodology oh the study
* To own a smartphone

Exclusion Criteria:

* Refusal to participate
* Patient on protective measures (guardianship or trusteeship)
* Deprived of liberty subject (administrative decision)
* Subject in exclusion period for another protocol
* Not affiliated to a social security agency
* Unable to understand and/or answer a questionnaire

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2018-05-31 (Actual); Primary Completion 2020-06-26 (Actual); Study Completion 2020-06-26 (Actual)

PRIMARY OUTCOMES:
Occurrence of a suicidal event during the follow-up | At 6 months
  Occurrence of a suicidal event will be checked by the Columbia Suicide Severity Rating Scale (C-SSRS) questionnaire and medical records at the end of study.

SECONDARY OUTCOMES:
Evaluation of the frequency of connection of the patient to the EMMA application | At 1 month
  The use is automatically measured by the application with the connection frequency
Evaluation of the frequency of connection of the patient to the EMMA application | At 2 months
  The use is automatically measured by the application with the connection frequency
Evaluation of the frequency of connection of the patient to the EMMA application | At 3 months
  The use is automatically measured by the application with the connection frequency
Evaluation of the frequency of connection of the patient to the EMMA application | At 4 months
  The use is automatically measured by the application with the connection frequency
Evaluation of the frequency of connection of the patient to the EMMA application | At 5 months
  The use is automatically measured by the application with the connection frequency
Evaluation of the frequency of connection of the patient to the EMMA application | At 6 months
  The use is automatically measured by the application with the connection frequency
Acceptability of EMMA assessed by the Smartphone application | At 1 month
  Questionnaire passed with the application (Likert scales)
Acceptability of EMMA assessed by the Smartphone application | At 2 months
  Questionnaire passed with the application (Likert scales)
Acceptability of EMMA assessed by the Smartphone application | At 3 months
  Questionnaire passed with the application (Likert scales)
Acceptability of EMMA assessed by the Smartphone application | At 4 months
  Questionnaire passed with the application (Likert scales)
Acceptability of EMMA assessed by the Smartphone application | At 5 months
  Questionnaire passed with the application (Likert scales)
Acceptability of EMMA assessed by the Smartphone application | At 6 months
  Questionnaire passed with the application (Likert scales)
Acceptability of EMMA assessed by the self assessment questionnaire Mobile Application Rating Scale (MARS) | At 6 months
Acceptability of EMMA assessed by a qualitative interview | At 6 months
  The qualitative interview is optional
Satisfaction of EMMA assessed by the Smartphone application | At 1 month
  Questionnaire passed with the application (Likert scales)
Satisfaction of EMMA assessed by the Smartphone application | At 2 months
  Questionnaire passed with the application (Likert scales)
Satisfaction of EMMA assessed by the Smartphone application | At 3 months
  Questionnaire passed with the application (Likert scales)
Satisfaction of EMMA assessed by the Smartphone application | At 4 months
  Questionnaire passed with the application (Likert scales)
Satisfaction of EMMA assessed by the Smartphone application | At 5 months
  Questionnaire passed with the application (Likert scales)
Satisfaction of EMMA assessed by the Smartphone application | At 6 months
  Questionnaire passed with the application (Likert scales)
Satisfaction of EMMA assessed by the satisfaction questionnaire | At 6 months
Satisfaction of EMMA assessed by a qualitative interview | At 6 months
  The qualitative interview is optional

CONTACTS AND LOCATIONS:
Locations (1):
- MontpellierUniversity Hopital, Montpellier, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Morgieve M, Genty C, Aze J, Dubois J, Leboyer M, Vaiva G, Berrouiguet S, Courtet P. A Digital Companion, the Emma App, for Ecological Momentary Assessment and Prevention of Suicide: Quantitative Case Series Study. JMIR Mhealth Uhealth. 2020 Oct 9;8(10):e15741. doi: 10.2196/15741. PMID 33034567